CLINICAL TRIAL: NCT03700840
Title: Interdental Microbiota According to the Caries Risk Factors Among Adolescents Aged 15 to 17 Years.
Brief Title: Interdental Microbiota Among Adolescents
Acronym: MIARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Montpellier (Other)
Collaborators: University of Lyon (Other)
Responsible Party: Principal Investigator, Paul TRAMINI, Ph.D. (department of public health), Université Montpellier
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-A00425-48
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Dental Caries; Gingivitis
Keywords: Oral biofilm; Microbiota; Adolescent; Dental carie
MeSH Terms: conditions — Dental Caries; Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical examination and sample (Other): Cross-sectional observational study
  Measure of 6 indices:
  * "Bleeding on Intergental Brush Index" (BOIB)
  * Gingivitis Score (GI)
  * Plaque index score (PI)
  * ICDAS
  * Salivary test
  Individual caries risk assessment
  Determination of interdental brushes adapted to each interdental site
  Recovery of the interdental brush passed through the 4 sites (between 15-16, 25-26, 35-36, 45-46) on which the interdental biofilm was fixed during the passage in the interdental space.
  The interdental brush is immediately put in a sterile tube and then sent in dry ice to maintain the integrity of the genetic material.
  Quantitative PCR experiments will be performed and a qualitative and quantitative analysis of the interdental flora will be made.
  Interventions: Device: Interdental brushes

INTERVENTIONS:
Device: Interdental brushes — interdental brush at 4 sites and PCR analysis

SUMMARY:
Adolescence remains a period during which tooth decay is still very active. There are few epidemiological studies in adolescents, and the majority of them were young people aged 15 and under. Early studies have characterized the interdental periodontal microbiota in healthy adults but, to our knowledge, no studies have analyzed the caries interdental microbiota in young people between 15 and 17 years of age. The main objective of this study is to describe the interdental microbiota in adolescents by a quantitative detection system using real-time PCR methodology. It will quantify 26 major interdental pathogens. The secondary objective is to analyse the distribution of these bacteria according to the level of caries risk and salivary risk.

Fifty Caucasian adolescents were recruited for this cross sectional study.

DETAILED DESCRIPTION:
Fifty Caucasian subjects were recruited from a pool of first-time volunteers who were referred to the Department of Public Health of the Faculty of Dentistry at the University of Montpellier, France. Written informed consent was obtained from all enrolled individuals in accordance with the Declaration of Helsinki. The study protocol was reviewed and approved by the Committee for the protection of persons (CPP) and by the National Commission of Informatics and Liberties, France.

Standardized clinical monitoring was performed 3 weeks before microbiological monitoring. The subjects were submitted to a medical/dental anamnesis, and information regarding their age, gender, and smoking status was obtained. The clinical examination was performed by trained and calibrated dentist. Clinical measurements were taken at six sites per tooth (mesio-buccal, buccal, disto-buccal, disto-lingual, lingual, and mesio-lingual) on all teeth, with the exception of the third molars, as previously described. The full-mouth clinical measurements included International Caries Detection and Assessment System (ICDAS), Caries Bleeding on interdental brushing index (BOIB), Gingival Index (GI), Plaque Index (PI) and Hygiene Index (HI), which were recorded on a dental chair, using a smooth probe, plane mirror and a surgical lamp.

Clinical assessments of the interdental spaces were performed using an IAP CURAPROX© colorimetric probe and registered the diameter of all the interproximal spaces of four pairs of teeth (premolar-molar). At the end of the examination visit, the participants were instructed to brush their teeth 3 h before the sampling visit and not to drink, eat or practice oral hygiene during this period.

In a group of 10 individuals who did not participate in this study, pairs of examinations were conducted in each individual, with a 1-h interval between them. Intraclass correlation coefficients for ICDAS, GI, PI, HI and BOIB were calculated at the site level. The intra- and inter-examiner coefficients for PI and HI ranged between 0.80 and 0.85, and between 0.75 and 0.85 for ICDAS.

For all subjects, the same four interdental sites (15-16, 25-26, 35-36, and 45-46) were assessed (total 200 sites). The appropriate prime interdental brushes were selected based on the clinical assessment of the interdental spaces.

With an alpha error of 5%, a power of 80%, an intraclass correlation coefficient of 0.8, a mean difference of bacteria counts between the 2 caries risk groups of 1,300,000, a total of 200 sites (which means 50 subjects) will be necessary.

Qualitative variables will be described by frequencies or percentages and quantitative variables by means and standard deviations. A Shapiro-Wilks test will be used to test the normality of the data. The comparison between the 2 caries risk groups will be achieved by a McNemar test for the qualitative variables and a Student test or a paired Wilcoxon test for the quantitative variables, depending on the normality of these variables.

The "clinical" questionnaire data completed by the dentist will be captured on a paper form provided at the beginning of the study. The forms thus recovered will be entered using a software to form the database. Paper forms will be archived with the study documents.

The bacteriological data obtained will be returned with the T envelope to the scientific manager and registered in the software.

The database created with the answers of "clinical" questionnaires and the results of the bacteriological analysis will be identified by order number and no surname data will be recorded on the electronic file thus created. At the end of the study, a report with the statistical tables and conclusions will be published for analysis and discussion of the data by the scientific committee and the project managers. Scientific publications will be written. The data is the property of the administrative manager of the study, no personal data will be released. Apart from the report and scientific publications, no data sharing is planned.

ELIGIBILITY:
Inclusion Criteria:

* presence of teeth 15-16-25-26-35-36-45-46
* At least of 22 teeth
* Good understanding of the French language
* One of the parents accepts the terms of the study and signs the written informed consent
* In good general health, without clinical abnormality and medical history
* Periodontal pocket greater than or equal to 3mm at interdental sites 15-16, 25-26, 35-36, 45-46

Exclusion Criteria:

* Smoking patient
* Patient with pathologies, orthodontic appliance
* Patient having taken antibiotics in the last 3 months
* Patient regularly using interdental brushes and / or dental floss and / or mouthwash
* Patient at risk for infectious endocarditis
* Patient unable to answer questions, non-cooperative

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of bacteria in the interdental plaque | through study completion, an average of 1 year
  Interdental sampling with a brush

SECONDARY OUTCOMES:
Distribution of bacteria according to different factors | through study completion, an average of 1 year
  Distribution of bacteria according to the level of caries risk, the salivary risk and other indices assessed during the clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Paul TRAMINI, PhD, Principal Investigator — paul.tramini@orange.fr
Locations (1):
- TRAMINI, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided